CLINICAL TRIAL: NCT06134908
Title: The Application of "Precise Education + Shared Decision-Making" Program for the Secondary Prevention of Fragility Fractures Based on Behavioral Theories: A Pilot Cluster Randomized Controlled Trial
Brief Title: PRevention of OsTEoporotiC FracTure 2 Pilot Study
Acronym: PROTECT-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); The Second Affiliated Hospital of Hunan University of Chinese Medicine (Unknown); Longgang Orthopedics Hospital of Shenzhen (Unknown); The First People's Hospital of Hefei (Other); Dongguan Eighth People's Hospital (Unknown); The Third People's Hospital of Longgang District Shenzhen (Unknown)
Responsible Party: Principal Investigator, Jian Mo, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PROTECT-2 Pilot
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Fragility Fracture
Keywords: Osteoporosis; Fragility Fracture; Shared Decision-Making; Education
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifaceted Intervention (Experimental): Group in the intervention arm will receive a multicomponent intervention at the clinician- and patient-level, with a shared decision-making booklet as well as a mobile application to promote osteoporosis management and fracture practice.
  Interventions: Behavioral: Multifaceted Intervention
- Usual-care Control (No Intervention): Group in the control arm will receive a leaflet and routine medical care per their existing health care providers.

INTERVENTIONS:
Behavioral: Multifaceted Intervention — The multicomponent intervention elements include education for clinicians and patients as well as a shared decision-making program among clinicians and patients. A shared decision-making booklet and a mobile application will be used to promote osteoporosis management and fracture practice.
  Arms: Multifaceted Intervention

SUMMARY:
With the aging of the world population, osteoporosis and fragility fractures have become global public health concerns. It has been estimated the population of people ≥60 years of age will increase from 229 million (16.2%) in 2017 to 479 million (35.1%) by 2050 in China. Because age is an important predictor of osteoporosis and fragility fracture, the incidence of fragility fracture has increased dramatically in China over the past decades. Timely treatment of osteoporosis is an effective way to decrease additional fracture risk among patients with fragility fractures, but anti-osteoporosis treatment rate is relatively low in China. Effective fracture prevention intervention is urgently needed in China.

As a potential way to achieve effective risk communication, shared decision-making allows patients to be active participants in the management of osteoporosis. The investigators designed a multifaceted intervention, which was named as "Precise Education + Shared Decision-Making" program for the secondary prevention of fragility fractures based on behavioral theories, and assessed the effectiveness for fracture prevention using a pilot cluster randomized controlled trial among several hospitals in China.

The aim of this pilot study is to test the acceptability and feasibility as well as preliminary efficacy of this program in patients with fragility fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Local residents (live in the city where the hospital is located for half a year or more);
2. Hospitalized patients with fractures aged 50 years and above;
3. First fracture, without history of fracture;
4. Never diagnosed as "osteoporosis" before admission;
5. No fracture history, and never receive any bone mineral density test, and never take anti-osteoporosis medication in the 4 years before admission;
6. Hospitalized patients with the following fractures: hip fracture, thoracic spine fracture, and lumbar spine fracture;
7. New fragility fracture: fracture that occurs after minor trauma or daily activities, such as a fracture caused by a fall from standing height or less; fracture happened within 6 weeks;
8. Not living in a nursing or rehabilitation institution before fracture;
9. Possess reading ability, and can read and understand informed consent forms or medical materials independently.

Exclusion Criteria:

1. Patients with pathological fractures caused by tumor or infection;
2. Patients with cognitive dysfunction or mental disorder;
3. AIDS patients;
4. Patients who refuse to follow-up, or have poor compliance for follow-up, or fail to understand and cooperate for follow-up;
5. Hearing or visual impairment, and unable to communicate or read materials;
6. Patients who have participate in other studies;
7. Other conditions that the investigator considered inappropriate to enroll.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility - Recruitment | 3 months
  Number or N (%) participants recruited within 3 months of trial initiation at each centre.
Trial feasibility - Acceptability of the multicomponent program component | 30 days after study recruitment
  Participants will be asked to evaluate the program with a questionnaire with questions about frequency, length, content, delivery, and duration of the booklet and the mobile application using a 5-point Likert scale.
Trial feasibility - Acceptability of the shared decision-making process | 7 days after study recruitment
  Both clinicians and patients will be asked to evaluate the shared decision-making process once they completed it. A survey will be administered to evaluate the content and comprehension of the program using a 5-point Likert scale.
Trial feasibility - Retention | 30 days after study recruitment
  The retention rates will be assessed as the 30-day follow-up rate.

SECONDARY OUTCOMES:
Anti-osteoporosis treatment rate | 1 month follow-up; 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  The patients will be followed up and asked whether they accept any anti-osteoporosis medication.
Shared decision-making process | 7 days after study recruitment
  Standardized questionnaires will be used to evaluated the shared decision-making process.
Bone mineral density test | 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  The patients will be followed up and asked whether they accept bone mineral density test.
Adherence of anti-osteoporosis medication | 1 month follow-up; 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  Adherence of anti-osteoporosis medication will be assessed with medication possession ratio and self-reported question.
Diagnosis, education, and follow-up practice of osteoporosis | 1 month follow-up; 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  The patients will be followed up with questionnaires about diagnosis, education, and follow-up of osteoporosis.
Refracture | 1 month follow-up; 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  The patients will be followed up and asked whether they have refracture.
Survival | 1 month follow-up; 3 month follow-up; 6 month follow-up; 12 month follow-up; 24 month follow-up
  The patients will be followed up about their survival status.
Patients' knowledge and attitude about osteoporosis and fragility fracture | baseline; 1 month follow-up; 6 month follow-up
  Patients' knowledge and attitude about osteoporosis and fragility fracture will be evaluated with standardized questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Mo, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Hunan University of Chinese Medicine, Changsha
  - Dongguan Eighth People's Hospital, Dongguan
  - Third Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First People's Hospital of Hefei, Hefei
  - Longgang Orthopedics Hospital of Shenzhen, Shenzhen
  - The Third People's Hospital of Longgang District Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No